CLINICAL TRIAL: NCT05969288
Title: Presence of Low Back Pain and Willingness to Osteopathic Cures in Italian Young People
Brief Title: Low Back Pain and Osteopathy in Italian Young People
Status: Recruiting | Type: Observational
Sponsor: International Institute of Behavioral Medicines (Other)
Responsible Party: Principal Investigator, Barbara Rocca, Scientific Director, International Institute of Behavioral Medicines
Other Study IDs: 2023-004
Record Dates: First submitted 2023-07-16; First posted 2023-08-01 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain
Keywords: Low back pain; Gnathology; Orthodontics; Osteopathy; Young people; Behavioral Medicine
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Behavioral survey — Behavioral survey by administering a short self-administered questionnaire (read more in the "Detailed description" section).

SUMMARY:
This is a behavioral observational study aimed at evaluating the presence of low back pain in young people and the intention to undertake osteopathic treatments. It consists of a short self-administered questionnaire which will be given to adolescents with gnathological/orthodontics disorders to complete. Relationships between low back pain of young individuals' answers with the intention to undertake osteopathic treatments will be evaluated.

DETAILED DESCRIPTION:
This is a behavioral observational study aimed at evaluating the presence of low back pain in young people and the intention to undertake osteopathic treatments.

Literature found out that low back pain is a common occurrence in young people. Adolescents develop frequently gnathological/orthodontics disorders. In Italy, young individuals with low back pain and gnathological/orthodontics disorders are frequently referred to osteopaths.

In Literature there are not studies which correlate low back pain, osteopathic cures and gnathological/orthodontics disorders as for young persons.

The study consists of a short self-administered questionnaire which will be given to young people to complete. In more details, the survey is made of 8 questions collecting information on presence/intensity of low back pain, intention to have osteopathic treatments, and (in that case) the satisfaction after the cures. Further, participants will have to complete a self-administered pain intensity numerical rating scale.

Descriptive statistics will be presented by taking into account the socio-demographic characteristics of the sample being investigated. Statistical correlations between adolescents' answers and the pain intensity numerical rating scale will be also evaluated.

This study investigates the relationships among low back pain, gnathological/orthodontics disorders, and osteopathic cures.

ELIGIBILITY:
Inclusion Criteria:

* common low back pain
* ability to read and understand the Italian language

Exclusion Criteria:

* any diagnosable cause of low back pain
* previous spinal surgery
* cognitive impairment
* refusal to adhere

Ages: 11 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Young people with low back pain and gnathological/orthodontics disorders.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
NRS | At the moment of the assessment
  Pain intensity Numerical Rating Scale: it a self-reported 11-point scale which evaluates pain intensity, varying from 0 (no pain at all) to 10 (the worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Rocca, Calosso, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salaffi F, Stancati A, Silvestri CA, Ciapetti A, Grassi W. Minimal clinically important changes in chronic musculoskeletal pain intensity measured on a numerical rating scale. Eur J Pain. 2004 Aug;8(4):283-91. doi: 10.1016/j.ejpain.2003.09.004. PMID 15207508
- [Result] Chiarotto A, Koes BW. Nonspecific Low Back Pain. N Engl J Med. 2022 May 5;386(18):1732-1740. doi: 10.1056/NEJMcp2032396. No abstract available. PMID 35507483